CLINICAL TRIAL: NCT06893341
Title: Monitoring Volatile Organic Compound Profiles in Exhaled Breath to Noninvasively Detect Glycemic Events in Patients With Diabetes
Brief Title: Monitoring Exhaled Breath to Noninvasively Detect Glycemic Events
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Mangilal Agarwal, Director, Integrated Nanosystems Development Institute, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22467
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Diabetes; Hyperglycemia; Hypoglycemia
Keywords: Volatile Organic Compound (VOC); Electronic Nose (e-Nose); Exhaled Breath; Noninvasive Health Monitoring
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Diabetic Children with Continuous Glucose Monitors (Experimental): These subjects will be given the Sensing Device, a wearable sensor that subjects can breathe into, which is being investigated in the current study as a potential medical device for noninvasive measurement of blood glucose.
  Interventions: Device: The Sensing Device

INTERVENTIONS:
Device: The Sensing Device — Children diagnosed with diabetes that wear a continuous glucose monitor will be given the Sensing Device. The subjects will provide breath samples into the device during euglycemia, hypoglycemia, and hyperglycemia, and the breath data will be analyzed to draw correlations with blood glucose levels.

SUMMARY:
The purpose of this study is to determine whether an array of biosensors can noninvasively identify hyperglycemic or hypoglycemic events in persons diagnosed with diabetes through noninvasive detection of volatile organic compounds in exhaled breath.

DETAILED DESCRIPTION:
A device has been developed for sensing volatile organic compounds (VOCs) from human breath. VOCs are chemicals in the air that make up scents and smells, and many VOCs are endogenously produced inside the human body. Trained dogs can smell exhaled breath to determine if someone has diabetes and can even distinguish hypo- or hyperglycemic events (low or high blood sugar). The purpose of this study is to determine if the sensor device can identify hypo- or hyperglycemic events in persons with diabetes through detecting VOCs in breath noninvasively. The data obtained from the VOC sensor will be compared to the information that is also gathered from a continuous glucose monitor (CGM) to establish correlations between blood glucose and exhaled VOC measurements.

ELIGIBILITY:
Inclusion Criteria:

* Who are diagnosed with type 1 diabetes.
* Who are between 12-19 years of age.
* That utilize a Dexcom (G6 or G7) continuous glucose monitoring device.
* That have an established working CGM for at least 12 hours (that does not need to be replaced within 24 hours).
* That are willing to share their daily CGM data for the study.
* That are the only individuals in their household with any type of diabetes diagnosis (type 1 or type 2).
* That are willing to return the device within 24-48 hours of study completion.
* That are located in Indianapolis, IN or its suburban areas.

Exclusion Criteria:

* That are smokers or use tobacco products or who live with someone who smokes in their vicinity.
* That have a condition or abnormality other than type 1 diabetes that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data.
* That utilize closed-loop diabetes management systems.
* That have symptoms or recently been diagnosed with an upper respiratory illness including COVID-19.
* That themselves or a close family member (living within the same household at the time of the data collection period) is on a "ketogenic diet".
* That themselves or a close family member is working in an industry with high and continuous exposure to exogenous VOCs. Examples of such industries include beauty salons and paint manufacturers.
* That are unable or unwilling to cooperate with sample collection.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between Breath Sensor Data and Blood Glucose | While wearing the device, up to 72 hours
  Participants will wear the breath sensor device for 72 hours. Participants will provide at least 15 direct breath samples during this time: one upon receipt of the device and in the presence of research staff, multiple during periods of hyperglycemia (blood glucose > 200 mg/dL), and multiple during periods of euglycemia. During each breath sample collection event, continuous CGM data will be recorded, and participants will also be asked to perform a finger-prick blood glucose test. Participants will return the device, and data from the wearable breath-based sensor will be analyzed using chemometrics and statistics to identify significant correlations between breath data and blood glucose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Linda A DiMeglio, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Only the principal investigators and research personnel listed in the approved Institutional Review Board (IRB) protocol will have access to the individual participant data (IPD), which will be stored on REDCap.

REFERENCES:
- [Background] Siegel AP, Daneshkhah A, Hardin DS, Shrestha S, Varahramyan K, Agarwal M. Analyzing breath samples of hypoglycemic events in type 1 diabetes patients: towards developing an alternative to diabetes alert dogs. J Breath Res. 2017 Jun 1;11(2):026007. doi: 10.1088/1752-7163/aa6ac6. PMID 28569238
- [Background] Woollam M, Angarita-Rivera P, Siegel AP, Kalra V, Kapoor R, Agarwal M. Exhaled VOCs can discriminate subjects with COVID-19 from healthy controls. J Breath Res. 2022 May 6;16(3). doi: 10.1088/1752-7163/ac696a. PMID 35453137
- [Background] Daneshkhah A, Shrestha S, Siegel A, Varahramyan K, Agarwal M. Cross-Selectivity Enhancement of Poly(vinylidene fluoride-hexafluoropropylene)-Based Sensor Arrays for Detecting Acetone and Ethanol. Sensors (Basel). 2017 Mar 15;17(3):595. doi: 10.3390/s17030595. PMID 28294961